CLINICAL TRIAL: NCT05265819
Title: Effect of Exergaming Exercises and Mediterranean Diet on Thyroid Cancer Patients Following Total Thyroidectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nabil Mahmoud Ismail Abdel-Aal (Other)
Responsible Party: Sponsor-Investigator, Nabil Mahmoud Ismail Abdel-Aal, Assistant Professor, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/003356
Record Dates: First submitted 2022-02-23; First posted 2022-03-04 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Diet, Mediterranean

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A (Active Comparator): Group A: Control group No intervention was provided for 12 weeks except thyroid hormone replacement therapy
  Interventions: Drug: thyroid hormone replacement therapy
- Group B (Experimental): Group B: Exergaming exercise The volunteers carried out 36 exergaming sessions
  Interventions: Device: X-BOX kinetic360
- Group C (Experimental): Group C: Mediterranean diet participants participated in the Mediterranean diet intervention for 12 weak and received dietary training from professional nutritionists at the baseline visit and samples of a Mediterranean diet for three times during the trial.
  Interventions: Dietary Supplement: mediterranean diet
- Group D (Experimental): Group D: Exergaming exercises and Mediterranean diet Exergaming exercises are used in addition to Mediterranean diet
  Interventions: Device: X-BOX kinetic360; Dietary Supplement: mediterranean diet

INTERVENTIONS:
Device: X-BOX kinetic360 — 1) Exergaming The practice of exergaming was performed using the Xbox 360 Kinect console,The volunteers carried out 36 exergaming sessions, with progressive increase in the duration of the games according to their tolerance,and reached a maximum duration of 50 minutes per session, included the realization of the games and the rest between activities. The exergaming protocol was performed two to three times a week, for a total of 12 weeks.
  Other Names: thyroid hormone replacement therapy
  Arms: Group B; Group D
Dietary Supplement: mediterranean diet — Mediterranean diet participants participated in the Mediterranean diet intervention for 12 weak and received dietary training from professional nutritionists at the baseline visit and samples of a Mediterranean diet for three times during the trial.
  Other Names: thyroid hormone replacement therapy
  Arms: Group C; Group D
Drug: thyroid hormone replacement therapy — thyroid hormone replacement therapy
  Arms: Group A

SUMMARY:
Effect of exergaming exercises and mediteranean diet on thyroid cancer patients following total thyroidectomy adult patients from both gender will be randomly assigned equally to exergaming exercises, Mediterranean diet groups using computer-generated block randomization.

Group A: Control group No intervention was provided for 12 weeks except thyroid hormone replacement therapy Group B: Exergaming exercise The volunteers carried out 36 exergaming sessions, with progressive increase in the duration of the games according to their tolerance,and reached a maximum duration of 50 minutes per session, included the realization of the games and the rest between activities. The exergaming protocol was performed three times a week, for a total of 12 weeks Group C: Mediterranean diet All participants participated in the Mediterranean diet intervention for 12 weak and received dietary training from professional nutritionists at the baseline visit and samples of a Mediterranean diet for three times during the trial.PREDIMED questionnaire is used To assess adherence to the Mediterranean diet Group D: Exergaming exercises and Mediterranean diet Exergaming exercises are used in addition to Mediterranean diet

DETAILED DESCRIPTION:
Outcome measures

1. Flow cytometry analyzer for NKC (CD3- CD16+ CD56+).
2. Immunoassay analyzer for thyroid profile (TSH,T3,T4)
3. Quality of life questionnaire
4. Fatigue questionnaire
5. PREDIMED questionnaire to asses diet adherence. Outcome measures will be measured at baseline and after 3 months of the treatement intervention

A) assessment

1. Quality of life questionnaire questionnaire
2. .Fatigue questionnaire
3. Adherence to diet A validated 14-item questionnaire for the assessment of adherence to the Mediterranean Diet (PREDIMED) will be recorded for all the enrolled subjects

   * Biochemical Analysis. [B] Intervention

     1. Exergaming The practice of exergaming was performed using the Xbox 360 Kinect console (Microsoft, Albuquerque, NM)
     2. Mediterranean diet All participants participated in the Mediterranean diet intervention for 12 weak and received dietary training from professional nutritionists at the baseline visit and samples of a Mediterranean diet for three times during the trial.

     4 groups will be randomly assigned Group A: Control group No intervention was provided for 12 weeks except thyroid hormone replacement therapy Group B: Exergaming exercise The volunteers carried out 36 exergaming sessions, with progressive increase in the duration of the games according to their tolerance,and reached a maximum duration of 50 minutes per session, included the realization of the games and the rest between activities. The exergaming protocol was performed three times a week, for a total of 12 weeks Group C: Mediterranean diet All participants participated in the Mediterranean diet intervention for 12 weak and received dietary training from professional nutritionists at the baseline visit and samples of a Mediterranean diet for three times during the trial.PREDIMED questionnaire is used To assess adherence to the Mediterranean diet Group D: Exergaming exercises and Mediterranean diet Exergaming exercises are used in addition to Mediterranean diet

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of thyroid papillary carcinoma as it is the most common type
2. Treatment with thyroid hormone medication after thyroidectomy
3. Lack of radioactive iodine treatment within the past 6 months
4. Blood hemoglobin level >10 g/dL.
5. Not taking drugs that could affect their immune function (e.g., immunosuppressants such as cyclosporin and steroids .
6. Lack of regular exercise
7. Age 18~45 years
8. Dose should be controlled at the first one year

   -

   Exclusion Criteria:

1) Abscess or inflammation suspected by preoperative tests 2) Patients with stage IV cancer and with limited understanding of assessment systems 3) History of head or neck malignancy . 4) Radiation therapy 5) Graves disease 6) Thyroiditis 7) Orthopaedic and rheumatic conditions of the neck . 8) The patient's inability to cooperate

-

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2022-12-05 (Estimated); Study Completion 2022-12-05 (Estimated)

PRIMARY OUTCOMES:
CD3- | 3 months
  CD3 (cluster of differentiation 3) is a protein complex and T cell co-receptor that is involved in activating both the cytotoxic T cell (CD8+ naive T cells) and T helper cells (CD4+ naive T cells). It is composed of four distinct chains.
  blood sample taken from the patients
CD16+ | 3 months
  CD16 is involved in antibody-dependent cell-mediated cytotoxicity and is expressed on large granular lymphocytes (LGLs) of both NK- and T-cell types.blood sample taken from the patients
CD56+ | 3 months
  CD56, is a member of the immunoglobulin superfamily engaged in both so-called homophilic and heterophilic interactions.blood sample taken from the patients

SECONDARY OUTCOMES:
TSH(thyroid stimulating hormone) | 3 months
  TSH stands for thyroid stimulating hormone. A TSH test is a blood test that measures this hormone.
T3 (triiodothyronine) | 3 months
  This test measures the level of triiodothyronine (T3) in your blood. T3 is one of two major hormones made by your thyroid
T4 (Thyroxine) | 3 months
  Thyroxine, also known as T4, is a type of thyroid hormone. This test measures the level of T4 in your blood. Too much or too little T4 can indicate thyroid disease.
Quality of life questionnaire | 3 months
  The World Health Organization (WHO) defined Quality of Life (QoL) as "an individual's perception of their position in life, in the context of the culture and value systems in which they live, and in relation to their goals, expectations, standards and concerns" . QoL is comprised of multiple aspects, including psychological health, physical well-being, social relationships, and environmental conditions [.
Fatigue questionnaire | 3 months
  questionnaire is applied to the patients

CONTACTS AND LOCATIONS:
Overall Officials: Mohsen Elsayyad, PhD, Study Director — Professor

IPD SHARING:
Plan to Share IPD: Yes
I will share my data
Supporting Information: Study Protocol, CSR
Time Frame: within 6 months of study completion
Access Criteria: It will be published in medical journals